CLINICAL TRIAL: NCT01017406
Title: PSU Heel Cushion for Treatment of Plantar Fasciitis:A Randomized Controlled Trial
Brief Title: Heel Cushion for Plantar Fasciitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Prince of Songkla University (Other)
Responsible Party: Boonsin Tangtrakulwanich, Department of Orthopedic Surgery, Faculty of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52-118-11-1-2
Record Dates: First submitted 2009-11-17; First posted 2009-11-20 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Plantar Fasciitis
Keywords: plantar fasciitis; heel cushion; treatment
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Plantar fascia stretching exercise (Experimental): Patient perform plantar fascia stretching 3 times per day
  Interventions: Device: PSU heel cushion and plantar fascia specific stretching exercise

INTERVENTIONS:
Device: PSU heel cushion and plantar fascia specific stretching exercise — * Wear heel cushion during daily activity
  * Plantar fascia stretching exercise 3 times per day

SUMMARY:
The investigators study aim to evaluate the efficacy of PSU heel cushion in treatment of plantar fasciitis. The investigators will do a randomized controlled trial in patient with plantar fasciitis compared with stretching exercise alone. The outcome measurement include heel pain improvement, compliance, satisfaction, foot functional score at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient with plantar fasciitis

Exclusion Criteria:

* Rheumatologic problem such as rheumatoid arthritis
* Latex allergy
* Pregnancy
* Previous surgery around foot and ankle

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
VAS score | 2 years

SECONDARY OUTCOMES:
Compliance | 2 years
Satisfaction score | 2 years
Foot functional score : FHSQ score | 2 years
Number of rescue pain killer | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Suntorn Wongsiri, MD., Principal Investigator — Department of orthopedic surgery, faculty of medicine
Locations (1):
- Prince of Songkla university, Hat Yai, Changwat Songkhla, Thailand